CLINICAL TRIAL: NCT06603441
Title: Reliability of the Samsung Galaxy for the Detection of Moderate to Severe Obstructive Sleep Apnea
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Principal Investigator, Robson Capasso, Professor of Otolaryngology - Head & Neck Surgery (OHNS), Stanford University
Other Study IDs: 76129
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Samsung Galaxy Watch technology: All participants screened will utilize the Samsung Galaxy Watch technology to monitor sleep patterns, oxygen saturation, PPG, and heart rate variability amongst other physiologic parameters. All data will be collected over the course of two intervention nights in the sleep lab and at home for three nights
  Interventions: Diagnostic Test: Samsung Galaxy Watch

INTERVENTIONS:
Diagnostic Test: Samsung Galaxy Watch — Samsung Galaxy Watch technology to monitor sleep patterns, oxygen saturation, PPG, and heart rate variability amongst other physiologic parameters.

SUMMARY:
The study will test the reliability of the Samsung Galaxy for the Detection of Moderate to Severe Obstructive Sleep Apnea (OSA)

DETAILED DESCRIPTION:
A prospective cohort of 150 individuals 22 years or older with a prior diagnosis or with a high likelihood of having moderate to severe OSA, screened using STOP-Bang and Epworth Sleepiness Scale questionnaires will be recruited and will utilize the Samsung Galaxy Watch technology to monitor sleep patterns, oxygen saturation, PPG, and heart rate variability amongst other physiologic parameters. All data will be collected over the course of two intervention nights in the sleep lab and at home for three nights.

ELIGIBILITY:
Inclusion Criteria:

* 22 years of age or older
* High pre-test likelihood of moderate to severe obstructive sleep apnea (OSA) based on screening questionnaires (STOP-Bang and Epworth Sleepiness Scale); or prior diagnosis of moderate-severe OSA.
* Able to provide informed consent confirmation

Exclusion Criteria:

* Severe and/or other acute medical illnesses as determined by the Investigator, in particular: Cardiac conditions such as Congestive Heart Failure (CHF), atrial fibrillation, Hx of Movement disorders: Parkinson's, Tremor, Lung conditions: Chronic Obstructive Pulmonary Disease (COPD), chronic bronchitis, emphysema, pulmonary fibrosis, acute episode of flu, allergies, asthma.
* Active comorbid sleep disorders, such as severe insomnia, restless legs syndrome, Periodic Leg Movement During Sleep (PLMS), narcolepsy, idiopathic hypersomnia
* Severe and/or unstable psychiatric disorders such as mood, anxiety, or psychotic disorders
* Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk
* Inability to use a Samsung Galaxy device for sleep tracking
* Inability to have two nights in the Stanford sleep lab.
* Participants who are pregnant
* Tattoos or scars covering the forearm area of both hands

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patient's visiting Stanford Hospital and Clinics
  2. Digital Recruitment - online advertisement campaign
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
4% Apnea Hypopnea Index (AHI) | Day 1 (Visit 1), Day 5 (Visit 2)
  Assessment of the 4% Apnea Hypopnea Index to determine the severity of sleep apnea

SECONDARY OUTCOMES:
User acceptance and feasibility of Galaxy Watch technology | Day 1 (Visit 1), Day 5 (Visit 2), At home monitoring (Day 2, 3 &4)
  Evaluation of,
  * Ease of use (scored from 1-5, where 1 indicates low ease of use and 5 indicates high ease of use)
  * Comfort (scored from 1-5, where 1 indicates low comfort and 5 indicates high comfort)
  * Compliance (dropout rate and the number of nights and hours of sleep recorded for each participant)

CONTACTS AND LOCATIONS:
Overall Officials: Robson Capasso, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided